CLINICAL TRIAL: NCT06252935
Title: A Single-Center, Evaluator-blind, Randomized Control Study to Assess the Effectiveness and Safety of Collagen Membrane (FormaAid®) in the Treatment of Periodontal Regeneration
Brief Title: Effectiveness and Safety of Collagen Membrane (FormaAid®) in the Treatment of Periodontal Regeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxigen Biotech Inc. (Industry)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBI-FA-202301
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Guided Tissue Regeneration; Collagen Membrane; Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FormaAid group (Experimental): Patients with intrabony defects are randomly assigned to receive either FormaAid collagen membrane or Geistlich Bio-Gide (control)before the GTR. And then treated with GTR surgery, the surgical procedure involves a full-thickness flap, the affected area is cleaned, and the damaged or diseased tissue may be removed. The allograft will be then placed into the defect and the collagen membrane is then trimmed and adapted over the defect. After all the treatment is done, 5-0 nylon suture will be used for the flap closure.
  Interventions: Device: FormaAid
- Bio-Gide group (Active Comparator): Patients with intrabony defects are randomly assigned to receive either FormaAid collagen membrane or Geistlich Bio-Gide (control)before the GTR. And then treated with GTR surgery, the surgical procedure involves a full-thickness flap, the affected area is cleaned, and the damaged or diseased tissue may be removed. The allograft will be then placed into the defect and the collagen membrane is then trimmed and adapted over the defect. After all the treatment is done, 5-0 nylon suture will be used for the flap closure.
  Interventions: Device: Bio-Gide

INTERVENTIONS:
Device: FormaAid — FormaAid is mainly composed of pure collagen extracted from bovine tendon, it is fabricated in the form of highly dense collagen matrix without chemical cross-linking to act as a barrier excluding epithelium.
  Arms: FormaAid group
Device: Bio-Gide — Bio-Gide is a bilayer collagen membrane made of porcine collagen, permits prompt and homogeneous vascularization and so brings about optimal tissue integration and wound stabilization.
  Arms: Bio-Gide group

SUMMARY:
The goal of this clinical trial is to evaluate clinically and radiographically effectiveness and products safety of the collagen membrane (FormaAid®) in the treatment of periodontal regeneration using guided tissue regeneration (GTR) performed by the trained periodontists. The main question it aims to answer are:

* The difference of periodontal status: clinical attachment level (CAL), periodontal pocket depth (PPD), gingival recession (GR), gingival Index (GI) and plaque index (PI).
* The difference of intrabony defect height.
* The difference of gingival tissue thickness and gingival tissue volume.
* The incidences of safety indicators.

Participants will be randomized into either experiment group or control group, undergo guided tissue regeneration (GTR) surgery at week 1, and re-visited on week 3, 5, 13 and 27 after the GTR surgery.

Researchers will compare if the test product is non-inferior to Bio-Gide.

DETAILED DESCRIPTION:
This study is conducted as a randomized controlled clinical trial regarding the use of two different marketed collagen membrane with freeze-dried bone allograft (FDBA) in treatment of periodontal intrabony defects. Collagen membrane acts as a barrier that prevents soft tissue (gums) from growing into the area where bone regeneration is desired. This allows the bone and other necessary tissues to regenerate more effectively. Sutures are removed 14 days after the surgery. Patients are then followed up at 5, 13- and 27-weeks post-surgery for Gl, PI, GR, PPD, and CAL to evaluate the tissue condition. The cone beam computed tomography (CBCT) and the X-ray radiographic evaluation will be assess in this study twice before and after treatment week 27 on the investigational site. And all subjects will receive intra-oral scanning with an intra-oral scanner at baseline and week 5, 13, 27 follow-up visits to assess the gingival tissue thickness and gingival tissue volume change. Safety data and adverse events would be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 70 years old, male or female
* Non current smoker: A person who has not smoked more than 100 cigarettes from the past to the present and has not smoked in the last 30 days.
* Patients who have decided to pay at their own expense and require guided tissue regeneration (GTR) for periodontal regeneration
* The defect morphology of intrabony defects is 2 or 3 wall intrabony defect.
* Periodontal pocket depth ≥ 5mm (probing periodontal depth, PPD, distance from gingival margin to the bottom of the defect).
* The height of the bone defect in the X ray image is ≥ 3mm (according to the X ray film intraosseous defect)
* The diagnosis of periodontal disease is stage III with either grade B or C.
* Patients who are willing to adhere to the study protocol and sign the informed consent form.
* Willing to accept evaluation during the trial period and return to clinic and treatment.
* Not a person subject to a sentence of guardianship or subject to judicial guardians.

Exclusion Criteria:

* Have a history of severe allergies or be allergic to collagen.
* Those who are known to be positive for human immunodeficiency virus.
* Poorly controlled diabetes (untreated or unstable disease status), blood test measurement of glycated hemoglobin greater than 7%
* Undergoing chemotherapy three months before agreeing to this experiment.
* Patients undergoing meat product desensitization treatment.
* Have a documented history of osteoporosis.
* Chronic disease, hypertension, hyperlipidemia, cardiovascular disease, and stroke not properly controlled (untreated or unstable disease condition) judged by the investigator at screening.
* Suffering from autoimmune diseases or connective tissue diseases, such as systemic lupus erythematosus or dermatomyositis.
* Coagulation disorder, lab test prothrombin time (PT) > 12 sec , or the use of anticoagulants that affects surgery judged by the investigator at screening.
* The tooth for which guided tissue regeneration (GTR) surgery is to be performed is determined to be furcation involved by investigator from image evaluation
* The tooth for which guided tissue regeneration (GTR) surgery is to be performed is considered unhealthy, exhibiting conditions such as apical lesion, needed endodontic therapy tooth, tooth fracture, etc. etc., as judged by the investigator f rom image evaluation
* Oral mucosal abnormalities or poor periodontal health, making it unsuitable for GTR surgical treatment, such as white spots, erythema, oral submucosal fibrosis, lichen planus, verrucous hyperplasia, inflammation, infection, etc. judged by the investigator at screening.
* Those whose periodontal cleaning is not in good condition or who are unable to cooperate with periodontal cleaning. Plaque control index (O'Leary index) >15%
* The mobility of the teeth that are to undergo guided tissue regeneration (GTR) surgery is greater than or equal to
* Teeth that are to undergo guided tissue regeneration (GTR) surgery have incomplete adjacent teeth on both sides, such as dental prostheses, crowns or bridges, artificial dental implants, or metal fillings. materials, etc., so as to affect the image evaluation.
* Others who are not suitable to participate in or continue this clinical trial as assessed by a physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference of clinical attachment level (CAL) | Week 0, Week 27
  Difference from baseline in periodontal clinical attachment level (CAL) with a periodontal probe Week 27 after the surgery. CAL is defined as periodontal probing depth plus gingival recession.

SECONDARY OUTCOMES:
Difference of periodontal pocket depth (PPD) | Week 0, Week 27
  PPD is assessed by periodontal probing to detect and measure the distance from gingival margin to the bottom of the defect. Difference from baseline in periodontal pocket depth (PPD) Week 27 after the surgery.
Difference of gingival recession (GR) | Week 0, Week 27
  GR is assessed by periodontal probing to detect and measure the distance from the gingival margin to the cemento-enamel junction (CEJ). Difference from baseline in periodontal Gingival recession (GR) Week 27 after the surgery.
Difference of gingival index (GI) | Week 0, Week 5, Week13, Week 27
  Difference from baseline in periodontal status: Gingival Index (GI) Week 5, 13, and 27 after the surgery. GI is evaluated according to Löe & Silness.
  * 0: Normal gingiva.
  * 1: Mild inflammation Slight change in color, slight oedema. No bleeding on probing.
  * 2: Moderate inflammation: Redness, oedema and glazing. Bleeding on probing.
  * 3: Severe inflammation: Marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.
Difference of plaque index (PI) | Week 0, Week 5, Week13, Week 27
  Difference from baseline in periodontal status: Plaque Index (PI) Week 5, 13, and 27 after the surgery. PI is evaluated by using the grading definition of Silness & Löe.
  * 0: No plaque in the gingival area.
  * 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth The plaque may only be recognized by running a probe across the tooth surface.
  * 2: Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  * 3: Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
Difference of intrabony defect height | Week 0, Week 27
  Difference from baseline in intrabony defect height (IDH) with X ray images Week 27 after the surgery. Bone Fill (%) is defined as the percentage change in IDH, following the equation: ((IDH week27 - IDH baseline)/ IDH baseline)*100%
Difference of gingival soft tissue | Week 0, Week 5, Week13, Week 27
  Difference from baseline in gingival soft tissue with an intra-oral scanning that gingival tissue thickness Week 5, 13, and 27 after the surgery. The baseline scanned data of all subjects would be superimposed with the corresponding scanned data obtained during re-evaluation to ensure the teeth are in the correct alignment and generate thickness change data.
Incidence of device related complications | Week 0 to Week 27
  The relationship of adverse events (AEs) to the investigational product will be assessed on four levels: highly probable, probable, possible, unlikely, and unrelated. The percentage of patients who experience AEs caused by the investigational product will be calculated to represent the incidence of device related complications.
Incidence of adverse event of special interest (AESI) / serious adverse event (SAE) | Week 0 to Week 27
  The incidence will be calculated to represent the percentage of patients who experience AESI or SAE. The AESI refer to specific adverse events in the GTR surgical site, including wound dehiscence, membrane exposure, wound infection, postoperative infection, operation site inflammation, pain, abscess, allergy, swelling and delayed healing. And the SAE is considered as adverse event that interrupt a subject's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually incapacitating.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-En Sung, Doctor, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No